CLINICAL TRIAL: NCT00795041
Title: Temporally Splitting Ovarian Stimulation and Embryo Transfer
Status: Completed | Type: Observational
Sponsor: University of Luebeck (Other)
Responsible Party: Buendgen N.; Griesinger G. PD Dr. med., University Hospital of SH, Campus Luebeck, Deparment of Obstetrics/Gynecology
Other Study IDs: TS1
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2008-11

CONDITIONS: Splitting of Ovarianstimulation and Embryotransfer
Keywords: vitrification; ovarian stimulation; reproductive medicine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: 10 women with indication for ART with ICSI or IVF

SUMMARY:
The purpose of this study is to explore the concept of temporally splitting ovarian stimulation and embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Indication for IVF/ICSI
* Age 18-36 years
* <= three earlier unsuccessful IVF/ICSI treatments with embryo transfer
* BMI 20-30
* Regular cycle with ovulation (28-35 days)
* Progesterone >7ng/ml at the beginning of stimulation
* Informed consents

Exclusion Criteria:

* PCOS (polycystic ovarian syndrome
* Endometrioses >= grade 3
* Known poor response syndrome
* History of ovariectomy
* Severe endocrinopathie

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women with indication for ART with ICSI or IVF
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-11; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | November 2008- May 2009

CONTACTS AND LOCATIONS:
Overall Officials: Georg Griesinger, PD MD, Principal Investigator — University of Schleswig-Holstein, Campus Luebeck, Department of Obstetrics and Gynecology
Locations (1):
- University Hospital of Schleswig Holstein, Campus Luebeck, Department of Obstetrics and Gynecology, Lübeck, Schleswig-Holstein, Germany

REFERENCES:
- [Derived] Buendgen NK, Schultze-Mosgau A, Cordes T, Diedrich K, Griesinger G. Initiation of ovarian stimulation independent of the menstrual cycle: a case-control study. Arch Gynecol Obstet. 2013 Oct;288(4):901-4. doi: 10.1007/s00404-013-2794-z. Epub 2013 Apr 3. PMID 23545834